CLINICAL TRIAL: NCT00734630
Title: A Randomized, Double-Blind, Placebo-Controlled Study of the Efficacy and Safety of Nebivolol Added To Antihypertensive Treatment With Lisinopril or Losartan in Patients With Hypertension.
Brief Title: Efficacy and Safety of Nebivolol (Added to Lisinopril or Losartan) in Hypertensive Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Noah Rosenberg , MD, Exec. Dir, Clin Dev, Cardiovascular and Metabolism, Forest Research Institute, a Subsidairy of Forest Laboratories, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NEB-MD-11
Record Dates: First submitted 2008-08-13; First posted 2008-08-14 (Estimated); Results first posted 2011-04-26 (Estimated); Last update posted 2011-04-26 (Estimated); Status verified 2011-03

CONDITIONS: Hypertension
Keywords: nebivolol; Bystolic ™; lisinopril; losartan; Hypertension
MeSH Terms: conditions — Hypertension | interventions — Nebivolol; Lisinopril

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nebivolol (Active Comparator): Nebivolol 5 mg, 5 mg nontrade tablets, oral administration Nebivolol 10 mg, 10 mg nontrade tablets, oral administration Nebivolol 20 mg, 20 mg nontrade tablets, oral administration Nebivolol 40 mg (two 20 mg nontrade tablets), oral administration
  Interventions: Drug: nebivolol
- Placebo (Placebo Comparator): Matching placebo tablets, oral administration
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: nebivolol — Encapsulated Nebivolol 5mg, 10mg, 20mg, or 40mg total daily dosage, oral administration once daily
  Lisinopril 10mg, 20mg total daily dosage, oral administration Losartan 50mg, 100mg total daily dosage, oral administration
  Other Names: Bystolic ™
  Arms: Nebivolol
Drug: Placebo — Lisinopril 10mg, 20mg total daily dosage, oral administration Losartan 50mg, 100mg total daily dosage, oral administration
  Other Names: Lisinopril-other names: Prinivil, Zestril; Losartan-other name: Cozaar
  Arms: Placebo

SUMMARY:
This study will assess blood pressure reduction with nebivolol or placebo in patients taking lisinopril or losartan.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, ambulatory outpatients 18-85 years old at screening
* Have a history of hypertension
* Qualifying laboratory results

Exclusion Criteria:

* Severe hypertension, including chronic kidney disease
* Documented congestive heart failure
* Have clinically significant respiratory, liver, or heart disease
* History of stroke, heart attack, or heart surgery in the last 6 months
* Have a history of hypersensitivity to nebivolol or other beta blockers.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 491 (Actual)
Dates: Start 2008-08; Primary Completion 2010-03 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manfred Stapff, MD, PhD, Study Director — Forest Research Institute, a subsidiary of Forest Laboratories, Inc.
Locations (75):
- United States (75):
  - Forest Investigative Site 070, Gulf Shores, Alabama
  - Forest Investigative Site 092, Huntsville, Alabama
  - Forest Investigative Site 058, Mesa, Arizona
  - Forest Investigative Site 059, Tempe, Arizona
  - Forest Investigative Site 024, Anaheim, California
  - Forest Investigative Site 012, Bell Gardens, California
  - Forest Investigative Site 026, Chino, California
  - Forest Investigative Site 083, Costa Mesa, California
  - Forest Investigative Site 030, Los Angeles, California
  - Forest Investigative Site 053, Orange, California
  - Forest Investigative Site 077, Riverside, California
  - Forest Investigative Site 034, Sacramento, California
  - Forest Investigative Site 028, Sacramento, California
  - Forest Investigative Site 048, San Bernardino, California
  - Forest Investigative Site 075, Santa Ana, California
  - Forest Investigative Site 087, Santa Ana, California
  - Forest Investigative Site 090, Temecula, California
  - Forest Investigative Site 010, Tustin, California
  - Forest Investigative Site 001, Westlake Village, California
  - Forest Investigative Site 061, Wheat Ridge, Colorado
  - Forest Investigative Site 046, Brooksville, Florida
  - Forest Investigative Site 015, DeLand, Florida
  - Forest Investigative Site 035, Fort Lauderdale, Florida
  - Forest Investigative Site 009, Hialeah, Florida
  - Forest Investigative Site 039, Hollywood, Florida
  - Forest Investigative Site 044, Jacksonville, Florida
  - Forest Investigative Site 002, Miami, Florida
  - Forest Investigative Site 085, Miami, Florida
  - Forest Investigative Site 091, Miami, Florida
  - Forest Investigative Site 013, Miami, Florida
  - Forest Investigative Site 052, Miami, Florida
  - Forest Investigative Site 049, Orlando, Florida
  - Forest Investigative Site 065, Pembroke Pines, Florida
  - Forest Investigative Site 041, Tampa, Florida
  - Forest Investigative Site 029, Atlanta, Georgia
  - Forest Investigative Site 068, Decatur, Georgia
  - Forest Investigative Site 050, Addison, Illinois
  - Forest Investigative Site 025, Chicago, Illinois
  - Forest Investigative Site 057, Chicago, Illinois
  - Forest Investigative Site 076, Joliet, Illinois
  - Forest Investigative Site 014, Orland Park, Illinois
  - Forest Investigative Site 079, Overland Park, Kansas
  - Forest Investigative Site 037, Auburn, Maine
  - Forest Investigative Site 045, Biddeford, Maine
  - Forest Investigative Site 003, Oxon Hill, Maryland
  - Forest Investigative Site 060, Prince Frederick, Maryland
  - Forest Investigative Site 042, Reisterstown, Maryland
  - Forest Investigative Site 023, Brockton, Massachusetts
  - Forest Investigative Site 066, Brockton, Massachusetts
  - Forest Investigative Site 040, Saint Clair Shores, Michigan
  - Forest Investigative Site 067, Rolling Fork, Mississippi
  - Forest Investigative Site 051, Edison, New Jersey
  - Forest Investigative Site 088, New York, New York
  - Forest Investigative Site 086, Syracuse, New York
  - Forest Investigative Site 006, Cary, North Carolina
  - Forest Investigative Site 022, Charlotte, North Carolina
  - Forest Investigative Site 064, Harrisburg, North Carolina
  - Forest Investigative Site 071, Raleigh, North Carolina
  - Forest Investigative Site 017, Wilmington, North Carolina
  - Forest Investigative Site 055, Fargo, North Dakota
  - Forest Investigative Site 007, Cincinnati, Ohio
  - Forest Investigative Site 054, Cleveland, Ohio
  - Forest Investigative Site 056, Perrysburg, Ohio
  - Forest Investigative Site 080, Ashland, Oregon
  - Forest Investigative Site 033, Eugene, Oregon
  - Forest Investigative Site 081, Harleysville, Pennsylvania
  - Forest Investigative Site 004, Greenville, South Carolina
  - Forest Investigative Site 031, Mt. Pleasant, South Carolina
  - Forest Investigative Site 018, Cleveland, Tennessee
  - Forest Investigative Site 043, Memphis, Tennessee
  - Forest Investigative Site 032, Nashville, Tennessee
  - Forest Investigative Site 008, Corpus Christi, Texas
  - Forest Investigative Site 063, San Antonio, Texas
  - Forest Investigative Site 062, San Antonio, Texas
  - Forest Investigative Site 016, Richmond, Virginia

REFERENCES:
- [Derived] Weiss RJ, Stapff M, Lin Y. Placebo effect and efficacy of nebivolol in patients with hypertension not controlled with lisinopril or losartan: a phase IV, randomized, placebo-controlled trial. Am J Cardiovasc Drugs. 2013 Apr;13(2):129-40. doi: 10.1007/s40256-013-0010-y. PMID 23519546

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occured from August 2008 through November 2009 at 76 US sites.
Pre-assignment Details: Placebo washout phase was required for patients currently on anti-hypertensives at screening followed by a losartan or lisinopril run-in phase before assignment to Placebo or Nebivolol arms. Patients who were untreated at screening started the study at the open-label lead-in phase.
Period: Overall Study
Arm/Group | Nebivolol | Placebo
Started | 258 | 233
Completed | 229 | 200
Not Completed | 29 | 33
Not completed — Lack of Efficacy | 4 | 4
Not completed — Withdrawal by Subject | 7 | 9
Not completed — Lost to Follow-up | 13 | 7
Not completed — Protocol Violation | 0 | 3
Not completed — Inclusion/Exclusion criteria not met | 0 | 1
Not completed — Adverse Event | 3 | 6
Not completed — Randomized in Error | 0 | 1
Not completed — Tested Positive for Illegal Drug Use | 1 | 1
Not completed — Poor Compliance | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nebivolol | Placebo | Total
Number analyzed (Participants) | 258 | 233 | 491
Age Continuous [Mean (Standard Deviation); unit: years] | 52.1 (10.1) | 53.8 (9.6) | 52.9 (9.9)
Age, Customized [Number; unit: Participants]
  Between 18 and 65 Years | 229 | 201 | 430
  ≥65 years | 29 | 32 | 61
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 104 | 92 | 196
  Male | 154 | 141 | 295
Region of Enrollment [Number; unit: participants]
  United States | 258 | 233 | 491

OUTCOME MEASURES:

1. Primary Outcome: Mean Seated Trough Cuff Systolic Blood Pressure (SBP) at Week 12
Description: Change from Baseline in Mean Seated Trough Cuff Systolic Blood Pressure (SBP) at Week 12, Last Observation Carried Forward (LOCF).
Time Frame: From baseline Visit 5 (Week 0) to Visit 10 (Week 12)
Measure: Mean (Standard Deviation); unit: mmHG
Arm/Group | Nebivolol | Placebo
Number analyzed (Participants) | 256 | 232
mmHG | -10.1 (16.9) | -7.3 (15.9)

2. Secondary Outcome: Mean Seated Trough Cuff Diastolic Blood Pressure (DBP) at Week 12
Description: Change from Baseline in Mean Seated Trough Cuff Diastolic Blood Pressure (DBP) at Week 12, Last Observation Carried Forward (LOCF).
Time Frame: From baseline Visit 5 (Week 0) to Visit 10 (Week 12)
Measure: Mean (Standard Deviation); unit: mmHG
Arm/Group | Nebivolol | Placebo
Number analyzed (Participants) | 256 | 232
mmHG | -7.8 (10.1) | -3.5 (10.6)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for a period of 21 months, from August 2008 to May 2010.
Description: 3 additional patients had a Serious Adverse Event(SAE), 1 instance of Coronary Artery Stenosis during the single-blind washout phase(SBWP), 1 instance of Myocardial Infarction during the open-label lead-in phase and 1 instance of deep vein thrombosis during the SBWP. The first 2 patients were not randomized. The 3rd patient was assigned placebo.
Arm/Group | Nebivolol | Placebo
Serious Adverse Events (participants affected / at risk) | 1/258 | 3/233
Other Adverse Events (participants affected / at risk) | 0/258 | 0/233
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nebivolol (N=258) | Placebo (N=233)
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Acute pancreatitis (Infections and infestations) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor can review results communications prior to public release & can embargo communications re: results for 60 days from time submitted to sponsor for review. PI shall not disclose sponsor's confidential information. Upon sponsor's request, PI shall delete any proprietary info & shall not include raw data in the publication. On sponsor's request, PI shall delay submission for any pub while sponsor files patent applications. Any publication will give recognition to Sponsor's support.